CLINICAL TRIAL: NCT01010659
Title: Prospective Clinical Evaluation of Dacryocystorhinostomy (DCR) With Lacrimal Intubation
Brief Title: The Safety and Efficacy of Lacrimal Silicone Intubation for the Management of Epiphora
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aurolab (Other)
Responsible Party: Dr. Usha Kim, Aravind Eye Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1PN1010940
Record Dates: First submitted 2009-11-05; First posted 2009-11-10 (Estimated); Last update posted 2011-07-15 (Estimated); Status verified 2011-07

CONDITIONS: Epiphora
Keywords: Dacryocystorhinostomy
MeSH Terms: conditions — Lacrimal Apparatus Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lacrimal Tube (Experimental): Dacryocystorhinostomy with silicone lacrimal intubation
  Interventions: Device: Lacrimal Tube

INTERVENTIONS:
Device: Lacrimal Tube — Lacrimal Tube
  Other Names: Auro-lac

SUMMARY:
The purpose of study is to investigate the safety and efficacy of lacrimal silicone intubation for the management of epiphora.

DETAILED DESCRIPTION:
Epiphora is an overflow of tears,usually caused by insufficient drainage of the tear film from the eye.The most common cause is a blockage of the lacrimal ducts located next to the nose, but the condition may also result from the excessive production of tears. Epiphora is a symptom rather than a disease and may be caused by a variety of conditions.

30 subjects will be recruited for this study, informed consent will be taken from the willing subjects. Complete ophthalmic evaluation would be performed including visual acuity. Diagnosis would be made on history of epiphora, regurgitation test, lids examination, nasal examination, probing and syringing. Standard procedure of Dacryocystorhinostomy (DCR) would be adopted in all cases with lacrimal intubation.

Syringing will be done on first follow up visit and skin sutures will also be removed. Tightness and mobility of the silicone tube will be checked. The tube is kept in place for 3-6 months according to need and then finally removed. The patency of lacrimal passage will be investigated by irrigation. A successful outcome will be defined as resolution of symptoms like epiphora and discharge and a patent lacrimal system on irrigation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects having epiphora
* Canalicular blockade ascertained with probing
* Chronic dacryocystitis
* Mucocele

Exclusion Criteria:

* Absent puncta
* Acute on chronic dacryocystitis
* Noticeable lid laxity
* Previous lacrimal surgery
* Patients younger than 15 years
* Suspicion of malignancy
* Post traumatic lids
* Bony deformity

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2009-11; Primary Completion 2011-03 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Resolution of epiphora | 15th Day, 1st Month, 6th Month and 12th month

SECONDARY OUTCOMES:
Post operative complications | 15th Day, 1st Month, 6th Month and 12th Month

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Usha Kim, MBBS, DO, Principal Investigator — Aravind Eye Hospital
Locations (1):
- Aravind Eye Hospital, Madurai, Tamil Nadu, India